CLINICAL TRIAL: NCT04434417
Title: Clinical Validation of a Simple and Fast Immunochromatographic Assay for Qualitative Determination of Specific ImmunoGLObulin IgG/IgM Antibodies to 2019- nCoV in Whole bLood, Serum or Plasma Specimen
Brief Title: Validation of an Immunochromatographic Assay for IgG/IgM Antibodies to 2019- nCoV
Acronym: I-GLOBAL
Status: Completed | Type: Observational
Sponsor: European Institute of Oncology (Other)
Collaborators: Azienda Socio Sanitaria Territoriale di Cremona (Other); Azienda Ospedaliera Niguarda Cà Granda (Other); Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); Papa Giovanni XXIII Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: I-GLOBAL
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: COVID
Keywords: immunoassay; immunoglobulin IgM; immunoglobulin IgG; cancer; COVID
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort tested: The cohort will include patients or health professionals who patients who were suspected of being infected with 2019-nCoV
  Interventions: Device: 2019-nCoV IgG/IgM Rapid Test Cassette

INTERVENTIONS:
Device: 2019-nCoV IgG/IgM Rapid Test Cassette — The specimen (whole blood, serum, plasma) will be loaded into the cassette and will migrate via capillary action along the membrane to react with the gold conjugate. The result will be available in 10 minutes

SUMMARY:
In COVID-19 pandemic, it is of critical importance to identify a rapid and simple diagnostic method to be used in clinical settings to timely inform and refine strategies that can prevent, control, and stop the spread of SARS-CoV-2. The 2019-nCoV IgG/IgM Rapid Test Cassette (Whole Blood/Serum/Plasma) is a qualitative, membrane-based immunoassay for the detection of immunoglobulin G (IgG) and Immunoglobulin M (IgM) antibodies to SARS-CoV-2 in whole blood, serum or plasma specimen. Clinical specimens from patients who were suspected of being infected with 2019-nCoV will be used to evaluate the performance of the assay.

DETAILED DESCRIPTION:
In COVID-19 pandemic, it is of critical importance to identify a rapid and simple diagnostic method to be used in clinical settings to timely inform and refine strategies that can prevent, control, and stop the spread of SARS-CoV-2. The 2019-nCoV IgG/IgM Rapid Test Cassette (Whole Blood/Serum/Plasma) is a qualitative, membrane-based immunoassay for the detection of Immunoglobulin G (IgG) and Immunoglobulin M (IgM) antibodies to SARS-CoV-2in whole blood, serum or plasma specimen. This test consists of two components, an IgG component and an IgM component. In the IgG component, anti-human IgG is coated in IgG test line region. During testing, the specimen reacts with 2019-nCoV antigen-coated particles in the test cassette. The mixture then migrates upward on the membrane chromatographically by capillary action and reacts with the anti-human IgG in IgG test line region, if the specimen contains IgG antibodies to SARS-CoV-2. The study aims to validate in a real life study a self diagnostic assay for SARS-CoV-2 with the advantages of high speed, simple operation and low cost, and overcomes the shortcomings of the existing molecular detection methods. Clinical specimens from patients who were suspected of being infected with 2019-nCoV will be used to evaluate the performance of the assay. In parallel, we will also use molecular assays for the detection of the presence of the viral RNA from nasopharyngeal swabs since Polymerase Chain Reaction is currently the gold standard.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected cases who meet the following 2 criteria at the same time:

   1. Epidemiological history: There was a history of contact with confirmed cases before the onset of illness; or subjects with at least one symptom in the last week before accrual in the trial. Subjects who have been in contact with people positive for SARS-CoV-2 in the previous 14 days.
   2. Clinical manifestations are defined as :

   Fever >37.5°; dry cough, muscle pain and/or fatigue, anosmia, subjects with respiratory distress (Respiratory Rate >25/min or O2 Saturation <92%) or imaging characteristics of pneumonia; or the total number of white blood cells is normal or decreased with the lymphocyte count decreased in the early stage of onset or there is an abnormal C-Reactive protein. Other symptoms that clinical investigator will relate to SARS-CoV-2 infection. Subject or cancer patients who have been quarantined for suspect symptoms and have access to hospital to continue therapy or to receive major surgery
2. Confirmed cases, namely patients or subjects with positive Reverse Transcription-Polymerase Chain Reaction (RT-PCR) for SARS-CoV-2. On the basis of meeting the criteria for suspected cases, sputum, throat swabs, lower respiratory tract secretions, and other specimens are tested by realtime RT-PCR for positive nucleic acid detection of new coronavirus; or viral gene sequencing is highly homologous with known new coronaviruses. Patients positive are serially tested with SARS-CoV-2 lgM / IgG Rapid Test to evaluate the immune response in IgG negative patients and the reliability of the test in those patients who develop clinical signs of SARS-CoV-2 during the trial.
3. Patients who are considered at high risk for infection and eligible for active therapy and major surgery

   * Frailty (age and multiple comorbidities) planned to receive a standard systemic anticancer treatment comprising chemotherapy and/or immunotherapy and/or radiation therapy or to receive an experimental treatment
   * Major surgery or surgery after neoadjuvant chemotherapy and or chemo/radiotherapy

Exclusion Criteria:

1. Ascertained influenza virus, parainfluenza virus, adenovirus, respiratory syncytial virus, rhinovirus, human metapneumovirus, Severe Acute Respiratory Syndrome coronavirus, and other known other viral pneumonia;
2. Ascertained mycoplasma pneumoniae, chlamydia pneumonia, and bacterial pneumonia; non-infectious diseases such as vasculitis, dermatomyositis, and organizing pneumonia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes:
  * Patients or health professionals already tested positive for the viral RNA from nasopharyngeal swabs by RT-PCR
  * Patients or health professional who are suspected of being infected with SARS-CoV-2 in the hospital
  * Patients who are considered at high risk for infection and eligible for active therapy and major surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the rate of SARS-CoV-2 positive cancer patients and health professionals in a comprehensive cancer center or in a cancer setting. | 6 months
  Patients positive are serially tested with SARSCoV-2 lgM / IgG Rapid Test to evaluate the immune response in IgG negative patients and the reliability of the test in those patients who develop clinical signs of SARS-CoV-2 during the trial.
Evaluation of test accuracy | 3 months
  The 2019-nCoV IgG/IgM Rapid Test Cassette (Whole Blood/Serum/Plasma) was compared with a leading commercial Polymerase Chain Reaction
Interleukin-6 quantification | 3 months
  Multiplex immunoassay
Interleukin-2 quantification | 3 months
  Multiplex immunoassay
Interleukin-1 quantification | 6 months
  Multiplex immunoassay
Tumor Necrosis Factor (TNF) quantification | 3 months
  Multiplex immunoassay
Interferon gamma quantification | 3 months
  Multiplex immunoassay

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Curigliano, MD, Principal Investigator — European IO; Antonio Marra, MD, Principal Investigator — European IO
Locations (5):
- Italy (5):
  - Papa Giovanni XXIII Hospital, Bergamo
  - Azienda Socio-Sanitaria Territoriale di Cremona, Cremona
  - European IO, Division of Early Drug Development for Innovative Therapies, Milan
  - Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta, Milan
  - Azienda Ospedaliera Niguarda Cà Granda, Milan

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available upon request
Supporting Information: Study Protocol, SAP, CSR
Time Frame: At the end of the study
Access Criteria: Upon request

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT04434417/Prot_SAP_000.pdf